CLINICAL TRIAL: NCT01323920
Title: Bortezomib-based Graft-Versus-Host-Disease Prophylaxis After Myeloablative Allogeneic Stem Cell Transplantation for Patients Lacking HLA-matched Related Donors: A Phase 2 Study
Brief Title: Bortezomib-based GVHD Prophylaxis After Allogeneic Transplant for Patients Without Matched Related Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-007
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndrome
Keywords: Stem Cell Transplant; Allogeneic Transplant; Donors
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes | interventions — Bortezomib; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade/Tac/MTX (Experimental): Drug: Bortezomib. Other Names: Velcade. Bortezomib 1.3 mg/m^2 IV
  Drug: Tacrolimus. Tacrolimus 0.05 mg/kg PO bid
  Drug: Methotrexate. Methotrexate 15 mg/m^2 IV
  Interventions: Drug: Bortezomib; Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.3 mg/m^2 IV
  Other Names: Velcade
Drug: Tacrolimus — Tacrolimus 0.05 mg/kg PO bid
Drug: Methotrexate — Methotrexate 15 mg/m^2 IV

SUMMARY:
A common problem after stem cell transplant is graft-versus-host-disease (GVHD). GVHD is a complication of transplantation where the donor graft attacks and damages some of your tissues. After stem cell transplant, all patients receive prophylactic medications against GVHD.

In this research study, we are studying the safety and effectiveness of a bortezomib based GVHD prophylaxic drug combination in participants after myeloablative allogeneic stem call transplantation from a matched unrelated donor, mismatched related or unrelated donor.

DETAILED DESCRIPTION:
Before your transplant you will receive conditioning therapy with fludarabine and busulfan given 7, 6, 5, and 4 days before your transplant. On day 0, you will receive selected blood cells taken from your sibling or unrelated donor.

You will receive 3 drugs for your GVHD prophylaxis:

Tacrolimus will be started 3 days before your transplant. It will be given intravenously and later by mouth. You will continue to take tacrolimus for 3 to 6 months after transplant.

Methotrexate will be given intravenously 1, 3, 6 and 11 days after your transplant.

Bortezomib will be given intravenously 1, 4, and 7 days after your transplant. On days 1, 4, 7, 30 and 3, 6 and 12 months after your transplant you will have a physical exam, blood work, and be asked to complete a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced and/or aggressive hematologic malignancy (including myelodysplastic syndrome) that is unlikely to be cured by alternative therapies
* HLA-Matched unrelated donor; or 1-locus HLA-mismatched related or unrelated donor
* ECOG performance status 0-2
* Adequate organ function
* Able to understand and willing to sign a written informed consent document
* Agrees to practice adequate contraception per study requirements

Exclusion Criteria:

* Pregnant or breastfeeding
* Recipient of prior allogeneic or autologous stem cell transplantation
* Prior abdominal radiation therapy
* HIV-positive on combination antiretroviral therapy
* Seropositive for hepatitis B or C
* Allergies to bortezomib, boron, or mannitol
* Myocardial infarction within last 6 months, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias
* Uncontrolled bacterial, viral or fungal infections
* Seizures or history of seizures
* History of another non-hematologic malignancy unless disease-free for at least 5 years
* Uncontrolled intercurrent illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MBBS, DPhil, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Koreth J, Kim HT, Lange PB, Bindra B, Reynolds CG, Chammas MJ, Armand P, Cutler CS, Ho VT, Glotzbecker B, Nikiforow S, Ritz J, Blazar BR, Soiffer RJ, Antin JH, Alyea EP 3rd. A Bortezomib-Based Regimen Offers Promising Survival and Graft-versus-Host Disease Prophylaxis in Myeloablative HLA-Mismatched and Unrelated Donor Transplantation: A Phase II Trial. Biol Blood Marrow Transplant. 2015 Nov;21(11):1907-13. doi: 10.1016/j.bbmt.2015.05.027. Epub 2015 Jun 6. PMID 26055298

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade/Tac/MTX: Drug: Bortezomib, Tacrolimus, Methotrexate
  Other Names:
  Velcade
  Bortezomib 1.3 mg/m^2 IV Tacrolimus 0.05 mg/kg PO bid Methotrexate 15 mg/m^2 IV
Period: Overall Study
Arm/Group | Velcade/Tac/MTX
Started | 35
Completed | 29
Not Completed | 6
Not completed — Death | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One participant signed consent and was enrolled onto study, however, was immediately taken off study because it became evident that the participant needed further therapy and was not ready to proceed to transplant.
Arm/Group | Velcade/Tac/MTX
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: The Cumulative Incidence of Grade II-IV Acute GVHD up to Day 100 After Stem Cell Infusion
Description: The primary outcome of this study is the cumulative incidence of grade II-IV acute GVHD up to Day 100 after stem cell infusion. Acute GHVD is graded according to the modified Glucksberg criteria (adapted from Thomas et al., NEJM ,1975, pp. 895-90), which is based on criteria by which the provider classifies acute GVHD per its objective organ staging. Acute GVHD is assessed in weekly standard of care visits post stem cell infusion and is captured in the protocol EDC upon evaluation of clinical notes up to Day 100. Data for acute GVHD organ staging and etiologies are collected in an acute GVHD separate case report form and do not include system organ class, expectedness or attribution.
Time Frame: Day 100
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade/Tac/MTX
Number analyzed (Participants) | 34
Percentage of participants | 32

2. Secondary Outcome: The Percentage Donor Engraftment up to Day 30 Post Stem Cell Infusion
Description: To assess the percentage donor engraftment up to day 30 post stem cell infusion, defined as the first of 3 consecutive days tested of documented absolute netrophil count (ANC) >/= 500 cells/u/L
Time Frame: Day 30
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade/Tac/MTX
Number analyzed (Participants) | 34
Percentage of participants | 94

3. Secondary Outcome: The Non-relapse Mortality, Progression-free and Overall Survival up to 1 Year After Stem Cell Infusion
Description: Progression free and overall survival by 1 year after stem cell infusion will be assessed using the method of Kaplan and Meier. Progression-free survival will be defined as the time from stem cell infusion to the time of disease progression or death from any cause. Overall survival will be defined as the time from stem cell infusion to the time to death from any cause. Patients will be censored at the time last documented alive. Cumulative incidence and Kaplan-Meier curves will be constructed as appropriate. Progression is defined per clinical presentation, not protocol specified, and vary per disease, e.g. blasts in bone marrow or peripheral blood for AML/MDS; lymphoma + on PET/CT re-staging etc.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number; unit: Percent of participants
Arm/Group | Velcade/Tac/MTX
Number analyzed (Participants) | 34
Percent of participants
  non-relapse mortality | 8.8
  progression-free survival | 85
  overall survival | 84

4. Secondary Outcome: The Cumulative Incidence of Chronic GVHD Requiring Systemic Immune Suppression up to 1 Year After Stem Cell Infusion
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Velcade/Tac/MTX
Number analyzed (Participants) | 34
Percentage of participants | 53

ADVERSE EVENTS:
Time Frame: All adverse events experienced by participants will be collected from the time of the first dose of study treatment, through the study and until the final study visit. Participants continuing to experience toxicity at the off study visit may be contacted for additional assessments until the toxicity has resolved or is deemed irreversible.Participants will be followed for 1 year after transplantation or until death, whichever occurs first.
Description: AEs grade 3-5 & SAEs whether reported by the participant, discovered during questioning, directly observed, or detected by physical examination, laboratory test or other means, will be recorded in the participant's medical record and on the appropriate study-specific case report forms. Participants removed from study treatment for unacceptable AEs will be followed until resolution or stabilization of the AE. One participant was enrolled but immediately taken off study for alternative therapy.
Arm/Group | Velcade/Tac/MTX
Serious Adverse Events (participants affected / at risk) | 5/34
Other Adverse Events (participants affected / at risk) | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade/Tac/MTX (N=34)
GVHD (Immune system disorders) | 2 (2) — 2 participants passed away to Grade 5 GVHD
HHV6/high LFTs (Infections and infestations) | 1 (1) — Grade 4 HHV-6 infection and elevated liver function tests
Sepsis (Infections and infestations) | 2 (2) — 2 participants passed away to Grade 5 sepsis
Relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Grade 5 AML relapse complicated by respiratory failure, B.O.S, and pneumonia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes